CLINICAL TRIAL: NCT03360097
Title: Pregnancy Outcomes in Patients With Slow Developing Blastocysts: What is the Best Transfer Strategy? A Prospective Randomized Controlled Trial
Brief Title: Clinical Outcomes of Slow Developing Blastocysts
Acronym: LATEBLOOM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants met the inclusion criteria in an exted period of time.
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Jorge Rodriguez-Purata, Principal Investigator, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMD-SLOW-2017-10
Record Dates: First submitted 2017-11-14; First posted 2017-12-02 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Infertility
Keywords: In vitro Fertilization; Slow Developing Blastocyst; Fresh Embryo Transfer; Frozen Embryo Transfer; Live Birth Rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: All participants will be randomized by an intention to treat approach. Randomization at the blastocyst stage is chosen to avoid cycle cancellation if randomized earlier. All components of the IVF/ICSI cycle including stimulation medications, monitoring protocols, etc. will be at the discretion of the participant's primary physician; while this information will be documented it will not constitute criteria for enrolment. The group allocation will take place the day of the embryo transfer. The clinician will randomize all included patients into one of the two study groups using an open computer-generated list. An interim analysis is planned and sample size will be plan accordingly, under the Pocok method, including 2 stages, with p-value as boundary scale, calculated to have 80% power to detect a 20% difference with a reference proportion of 25% clinical pregnancy rate and a one-sided (upper) alpha of 0.025
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh ET (No Intervention): The best available embryo is at expansion grade <4 by Gardner classification 5 days after oocyte retrieval. Patient's embryos are cultured to day 6 and transferred regardless of expansion grade. Arrested blastocysts are discarded.
- Frozen Embryo Transfer (Experimental): The best available embryo is at expansion grade <4 by Gardner classification 5 days after oocyte retrieval. Patient's embryos are cultured to day 6 and vitrified regardless of expansion grade. Arrested blastocysts are discarded. The single best available embryo is transferred under a cryo-synthetic cycle.
  Interventions: Procedure: Frozen Embryo Transfer

INTERVENTIONS:
Procedure: Frozen Embryo Transfer — Patient's embryos are cultured to day 6, vitrified and transferred in a cryo-synthetic cycle
  Arms: Frozen Embryo Transfer

SUMMARY:
This study evaluates which transfer strategy will result in a higher probability of pregnancy in patients whose single best day 5 embryo resulting from an IVF cycle is classified as expansion grade <4 by Gardner and Schoolcraft classification. All cycles will be cultured to day 6 and half the patients will undergo a fresh embryo transfer and the other half a frozen embryo transfer.

DETAILED DESCRIPTION:
A lack of established markers for predicting blastocyst development increases the risk of having no embryos or embryos not-fully expanded available for transfer. Slower but non-arrested embryos are frequently found to have progressed to blastocyst stage by the time of a day 6 transfer. In the absence of a receptive endometrium, embryo selection for fresh transfer may be futile, and cryopreservation could be a better option. The objective is to determine which transfer strategy will result in a higher probability of pregnancy in patients whose single best day 5 embryo resulting from an IVF cycle is classified as expansion grade <4 by Gardner and Schoolcraft classification. The investigators hypothesize that in bad prognosis patients with slow-developing blastocysts, vitrified-warmed embryo transfer will result in higher implantation, clinical and ongoing pregnancy and live birth rates than fresh embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* All IVF cycles undergoing autologous fresh blastocyst embryo transfer
* All IVF cycles in which the best available embryo for transfer is at expansion grade <4
* All ages

Exclusion Criteria:

* Ovum Donation cycles
* Preimplantation genetic testing cycles

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 20 days after date of embryo transfer
  Proportion of patients with the presence of a gestational sac seen by transvaginal ultrasonography 20 days after the embryo transfer

SECONDARY OUTCOMES:
Biochemical Pregnancy Rate | 9 days after date of embryo transfer
  Proportion of patients with the detection of β-hCG level ≥5 mIU/mL 9 days after the embryo transfer
Live Birth Rate | 24 weeks after the embryo transfer
  Proportion of patients which deliver a live infant after 24 weeks of gestation
Miscarriage Rate | 14 weeks after the embryo transfer
  Proportion of patients with a pregnancy loss following a positive pregnancy test and/or detectable gestacional sac
Cryopreservation-thaw rate | 1 day after the thawing procedure
  Proportion of vitrified blastocysts which survive the re-warming

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Rodriguez-Purata, MD, Principal Investigator — Fundacion Dexeus
Locations (1):
- Institut Universitari Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2020
Access Criteria: All